CLINICAL TRIAL: NCT00525083
Title: Protein and Phospholipid Analysis of HDL in Patients With Very High Serum Levels of HDL-C
Status: Terminated | Type: Observational
Why Stopped: PI left for another institution
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 050806
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hyperlipidemia
Keywords: hyperlipidemia; HDL-C; low density lipoprotein
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, HDL preps, genomic DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary heart disease (CHD) is the single leading cause of death in the United States . Serum Cholesterol is known to have a direct impact on a number of human diseases through a variety of mechanisms. This is particularly true of cardiovascular disease. Measurement and manipulation of serum cholesterol has become a primary focus of primary care physicians and cardiologists when attempting to reduce risk of heart disease.

DETAILED DESCRIPTION:
Clinical investigations have shown that lowering the "total serum cholesterol" levels result in a significant reduction of coronary artery disease and myocardial infarctions . Thus, interventions to lower the "total serum cholesterol" are commonly employed by medical professionals - this includes behavioral modifications (exercise, dieting, and weight loss) and pharmacological interventions.

Investigation has shown that clinical outcomes do not only rely on "total serum cholesterol". "Total serum cholesterol" is comprised of multiple subtypes - most notable are "HDL Cholesterol" and "LDL cholesterol". Analysis of the data has shown that high levels of LDL cholesterol predict higher rates of cardiovascular events, while high levels of HDL cholesterol are actually predictive of significantly less cardiovascular events. These effects are independent of other cardiovascular risk factors .

The mechanism by which LDL cholesterol results in heart disease has been intensely investigated and elucidated. Numerous drugs are now approved and utilized by physicians to lower the LDL cholesterol of patients to prevent primary and secondary cardiovascular disease.

Epidemiological data show that low levels of HDL-C place individuals at higher risk for coronary artery disease while high levels of HDL-C actually decrease an individual's risk . The mechanism behind this risk reduction remains unclear and is likely multi-factorial. Furthermore, some data suggests that while HDL-C is important in risk reduction, it is not necessarily the measured serum level of HDL-C, but also the composition, oxidation state, metabolism of the HDL-C that determines an individual's cardiac risk . Understanding of this mechanism could lead to potential therapeutic targets as well as clinically relevant diagnostic testing.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Serum HDL-C > 100 mg/dL.

Exclusion Criteria:

* Significant history of smoking.
* Diabetes Mellitus.
* Severe hypertension.
* Age > 65 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HDL above 100 mg/dl and with personal or family history of early atherosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2014-11-03 (Actual); Study Completion 2014-11-03 (Actual)

PRIMARY OUTCOMES:
Identification of protein or phospholipid signature suggestive of dysfunctional HDL | 2013-2016

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Fazio, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States